CLINICAL TRIAL: NCT02326090
Title: A Phase 2, Multi-Center, Randomized, Double Masked, Placebo Controlled Clinical Study to Assess the Safety and Efficacy of 1.0% and 2.5% Cis-UCA Ophthalmic Solutions in Subjects With Dry Eye
Brief Title: Phase 2 Study With Cis-UCA Ophthalmic Solutions in Subjects With Dry Eye
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herantis Pharma Plc. (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL12002 / 14-110-0005
Record Dates: First submitted 2014-12-22; First posted 2014-12-25 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- cis-UCA ophthalmic solution 1.0% (Active Comparator): One drop in each eye
  Interventions: Drug: cis-UCA ophthalmic solution 1.0%
- cis-UCA ophthalmic solution 2.5% (Active Comparator): One drop in each eye
  Interventions: Drug: cis-UCA ophthalmic solution 2.5%
- Placebo ophthalmic solution (Placebo Comparator): One drop in each eye
  Interventions: Drug: Placebo ophthalmic solution

INTERVENTIONS:
Drug: cis-UCA ophthalmic solution 1.0%
  Arms: cis-UCA ophthalmic solution 1.0%
Drug: cis-UCA ophthalmic solution 2.5%
  Arms: cis-UCA ophthalmic solution 2.5%
Drug: Placebo ophthalmic solution
  Arms: Placebo ophthalmic solution

SUMMARY:
The objective of the Phase 2 study is to compare the safety and efficacy of cis-UCA Ophthalmic Solutions to placebo for the treatment of the signs and symptoms of dry eye.

ELIGIBILITY:
Key Inclusion Criteria:

* Be at least 18 years of age;
* Provide written informed consent;
* Have a subject reported history of dry eye;
* Have a history of use or desire to use eye drops.

Key Exclusion Criteria:

* Have any clinically significant eye findings that require therapeutic treatment, and/or in the opinion of the Investigator may interfere with study parameters;
* Have worn contact lenses within 7 days of Visit 1 or anticipate using contact lenses during the study;
* Have previously had laser-assisted in situ keratomileusis (LASIK) surgery within the last 12 months;
* Have used Restasis® within 30 days of Visit 1;
* Have any planned ocular and/or lid surgeries over the study period;
* Be a woman who is pregnant, nursing or planning a pregnancy;
* Be unwilling to submit a urine pregnancy test at Visit 1 and Visit 4 (or early termination visit) if of childbearing potential;
* Have a known allergy and/or sensitivity to the study drug or its components;
* Have a condition or be in a situation which the Investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study;
* Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days of Visit 1;
* Be unable or unwilling to follow instructions, including participation in all study assessments and visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2014-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Corneal Fluorescein Staining | Day 29
Symptom Score | Day 22 to 28

CONTACTS AND LOCATIONS:
Locations (1):
- Andover, Massachusetts, United States